CLINICAL TRIAL: NCT02749656
Title: A Randomized Control Trial of Efficacy and Safety of 0.25% Desoximetasone Cream (Topoxy®) Compared With 0.25% Desoximetasone Cream (Topicorte®) in the Treatment of Scalp Psoriasis
Brief Title: Efficacy and Safety of 0.25% Desoximetasone Cream (Topoxy®) in the Treatment of Scalp Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Collaborators: SPS MEDICAL CO.,LTD. (Unknown); Siriraj clinical research center (Unknown)
Responsible Party: Principal Investigator, Pichanee Chaweekulrat, M.D., Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPS01
Record Dates: First submitted 2016-04-19; First posted 2016-04-25 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Scalp Psoriasis
Keywords: Scalp psoriasis; 0.25% Desoximetasone cream
MeSH Terms: interventions — Desoximetasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.25% Desoximetasone cream (Topoxy®) (Experimental): 0.25% Desoximetasone cream (Topoxy®): apply on scalp psoriasis lesion twice a day for 8 weeks.
  (Tar shampoo will be given to all participants. The Shampoo should be applied on wet scalp every other day, then massage and allow shampoo to remain on the scalp for 5 minutes, after that rinse off by water.)
  Interventions: Drug: 0.25% Desoximetasone cream (Topoxy®)
- 0.25% Desoximetasone cream (Topicorte®) (Active Comparator): 0.25% Desoximetasone cream (Topicorte®): apply on scalp psoriasis lesion twice a day for 8 weeks.
  (Tar shampoo will be given to all participants. The Shampoo should be applied on wet scalp every other day, then massage and allow shampoo to remain on the scalp for 5 minutes, after that rinse off by water.)
  Interventions: Drug: 0.25% Desoximetasone cream (Topicorte®)
- Placebo (Placebo Comparator): Placebo: apply on scalp psoriasis lesion twice a day for 8 weeks. (Tar shampoo will be given to all participants. The Shampoo should be applied on wet scalp every other day, then massage and allow shampoo to remain on the scalp for 5 minutes, after that rinse off by water.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.25% Desoximetasone cream (Topoxy®) — apply on the scalp psoriasis lesion twice a day
  Other Names: Topoxy®
  Arms: 0.25% Desoximetasone cream (Topoxy®)
Drug: 0.25% Desoximetasone cream (Topicorte®) — apply on the scalp psoriasis lesion twice a day
  Other Names: Topicorte®
  Arms: 0.25% Desoximetasone cream (Topicorte®)
Drug: Placebo — apply on the scalp psoriasis lesion twice a day
  Other Names: vehicle
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of 0.25% Desoximetasone cream (Topoxy®) compare with 0.25% Desoximetasone cream (Topicorte®) in the treatment of scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosed with scalp psoriasis by dermatologist
3. Has scalp psoriasis Involve ≥ 10% of total scalp area and also has clinical signs, or a previous diagnosis, of psoriasis on the trunk and/or limbs
4. Total severity of scalp psoriasis should be graded in mild to very severe according to Investigator's Global Assessment score (IGA)
5. Clinical signs (redness, thickness, scaliness) should be scored as "Moderate" for at least 1 sign and "slight" on each of the other two signs
6. All participants agree to participate in the study and already complete and sign consent form

Exclusion Criteria:

1. Treated with these medications before including in the study

   * Topical corticosteroid for scalp psoriasis (except emollients and shampoo) within 2 weeks
   * Very potent topical corticosteroids for psoriasis on other area or Narrow band Ultraviolet B (NB-UVB) within 2 weeks
   * Oral psoralen plus Ultraviolet A (PUVA) or oral medication (Methotrexate, Acitretin, Cyclosporine) within 4 weeks
   * Biologic agents or concomitant medication that could affect scalp psoriasis (Beta- blockers, Antimalarial drugs, Lithium ) within 6 months
2. Has skin infection or atrophic skin on the scalp
3. Has history of allergic reaction or hypersensitivity to 0.25% Desoximetasone
4. Female participants with pregnancy or in lactation period
5. Participants who unable to come for follow-up visits at hospital
6. Participants with other underlying disease e.g. diabetes mellitus, hypertension, thyroid disease
7. Vulnerable subject e.g. illiterate person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of Investigator's Global Assessment score (IGA) after treatment | 2, 4 and 8 weeks
  The Investigator's Global Assessment score (IGA) was recorded at the first visit and after treated 2,4 and 8 weeks with 0.25% Desoximetasone cream (Topoxy®), 0.25% Desoximetasone cream (Topicorte®) or placebo. The IGA score consisted of 6 points score (0 = absent disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, 4 = severe disease and 5 = very severe disease)

SECONDARY OUTCOMES:
Change of total sign score (TSS) after treatment | 2, 4 and 8 weeks
  The Total sign score (TSS) was recorded at the first visit and after treated 2,4 and 8 weeks with 0.25% Desoximetasone cream (Topoxy®), 0.25% Desoximetasone cream (Topicorte®) or placebo. The TSS score was the sum of 5-point rating scores for erythema, induration and scaling (0 = no sign, 1 = slight signs, 2 = moderate signs, 3 = severe signs and 4 = very severe signs)
Number of patients with clear or absent disease after treatment | 8 weeks
  Number of patients with clear or absent disease were recorded after treated 8 weeks with 0.25% Desoximetasone cream (Topoxy®), 0.25% Desoximetasone cream (Topicorte®) or placebo.
Side effects after treatment | 2, 4 and 8 weeks
  Cutaneous side effects (e.g. skin discomfort, skin atrophy, telangiectasia) from 0.25% Desoximetasone cream were recorded after treated 2, 4 and 8 weeks.
  The side effects were scored as 0 = none, 1 = mild, 2 = moderate, 3 = severe for skin discomfort, skin atrophy and telangiectasia.

CONTACTS AND LOCATIONS:
Overall Officials: Associated. Prof. Chanisada Wongpraparut, M.D., Principal Investigator — Mahidol University; Assist. Prof. Leena Chularojmontri, M.D., Study Chair — Mahidol University; Assist. Prof. Narumol Silpa-archa, M.D., Study Chair — Mahidol University; Pichanee Chaweekulrat, M.D., Study Chair — Mahidol University
Locations (1):
- Department of dermatology Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kircik L, Lebwohl MG, Del Rosso JQ, Bagel J, Stein Gold L, Weiss JS. Clinical study results of desoximetasone spray, 0.25% in moderate to severe plaque psoriasis. J Drugs Dermatol. 2013 Dec;12(12):1404-10. PMID 24301242
- [Background] Kuokkanen K. Comparison of 0.25% desoxymethasone ointment with 0.05% fluocinonide ointment in psoriasis. Curr Med Res Opin. 1976-1977;4(10):703-5. doi: 10.1185/03007997609112005. PMID 800971